CLINICAL TRIAL: NCT04272294
Title: Functional and Molecular Characterization of Treatment Response in Tumors in the Oral Cavity Using Optical Spectroscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never initiated
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 239327
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Spectrum Analysis, Raman

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Use of Optical Spectroscopy (Experimental): Optical spectroscopy used to characterize treatment response
  Interventions: Device: Optical Spectroscopy

INTERVENTIONS:
Device: Optical Spectroscopy — Using oral spectroscopy device to characterize treatment response in tumors

SUMMARY:
The objective of this pilot study is to estimate the sensitivity and specificity of diffuse reflectance spectroscopy (DRS) and Raman spectroscopy (RS) at detecting treatment-resistant disease when DRS and RS are used together to measure treatment-induced reoxygenation and molecular changes in tumors of the oral cavity. This study will be performed in a total of 90 patients that have Stage 3 or 4 head and neck squamous cell carcinoma (HNSCC) with primary tumors located in the larynx or one tonsil.

DETAILED DESCRIPTION:
The objective of this pilot study is to estimate the sensitivity and specificity of diffuse reflectance spectroscopy (DRS) and Raman spectroscopy (RS) at detecting treatment-resistant disease when DRS and RS are used together to measure treatment-induced reoxygenation and molecular changes in tumors of the oral cavity. This study will be performed in a total of 90 patients that have Stage 3 or 4 head and neck squamous cell carcinoma (HNSCC) with primary tumors located in the larynx or one tonsil.

This study is a single-arm, single-center observational pilot study of the accuracy of DRS+RS at distinguishing early between treatment-resistant and treatment-responsive disease in study-eligible subjects undergoing first-line chemoradiation therapy for Stage 3 or 4 HNSCC of the larynx or tonsil.

Three (3) optical spectra each will be collected from the tumor, an adjacent normal site, and a normal tissue site on the buccal mucosa prior to treatment. The subject will undergo 4 repeat post-treatment measures taken after radiation therapy begins (marked as Day 1). Repeat measures will be taken on Day 2(+1), Day 4(±1), Day 7(±1), and Day 10(±1). The probe will be performed at the beginning of the radiation therapy visit, prior to the radiation dose that day.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of stage 3 or 4 HNSCC with documentation of HPV status
* Tumor located in one of the tonsils and/or larynx
* Expected to have ability to tolerate laryngoscope procedure
* Must sign Informed Consent Form
* Scheduled for chemoradiation therapy

Exclusion Criteria:

* Previous oral cavity or tonsil or pharyngeal surgery or therapy related to the disease
* Disease in both tonsils
* Patients who, in opinion of Investigator, should not participate
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Successful identification of treatment-resistant disease | 3 weeks
  a sensitivity estimate of 70%, i.e., successful identification of treatment-resistant disease in 70% of the patients who have it (as defined by RECIST v1.1) before Week 3 of treatment will constitute a benchmark of success.

CONTACTS AND LOCATIONS:
Overall Officials: Moreno Mauricio, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No